CLINICAL TRIAL: NCT06410742
Title: Exploring the Role of Central Sensitization on Biopsychosocial Factors in Primary Sjögren's Syndrome: a Cross-Sectional Analysis
Brief Title: The Role of Central Sensitization on Biopsychosocial Factors in Primary Sjögren's Syndrome
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Nazli Elif Nacar, Lecturer, Kahramanmaras Sutcu Imam University
Other Study IDs: Kahramanmaras.SU
Record Dates: First submitted 2024-05-06; First posted 2024-05-13 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-12

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren' Syndrome; correlation; xerostomia; dryness
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with primer Sjogren's syndrome

SUMMARY:
Following the guidance of individuals with primary Sjögren's Syndrome who receive diagnosis, routine medical care, and treatment management, the evaluations will be performed once by the researchers and will take approximately one hour.

In addition, healthy individuals with a similar average age to the evaluation group without any disease diagnosis will be included in the study as a control group. Evaluations of the healthy group will be made once by the researchers and will take approximately one hour.

Data will be collected face to face at the Faculty of Physical Therapy and Rehabilitation, Rheumatology Unit.

Data collection tool of the research:

* Information about patients will be recorded with the Demographic Information Form.
* EULAR Sjögren's Syndrome Disease Activity Index
* EULAR Sjögren's Syndrome Patient Reporting Index
* Primary Sjögren's Syndrome Quality of Life Scale
* BETY-Biopsychosocial Questionnaire
* Central Sensitization Scale
* Pain Catastrophizing Scale
* Hospital Anxiety and Depression Scale
* Multidimensional Fatigue Rating Scale
* Turkish Eating Assessment Tool
* Yale Swallow Protocol
* Test of Mastication and Swallowing Solids
* Dysphagia Limit Test
* Xerostomia inventory

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Primary Sjögren's Syndrome
* 18 years or older

Exclusion Criteria:

* Patients with Secondary Sjögren's Syndrome,
* Patients who are diagnosed with other uncontrolled/clinically important diseases (chronic obstructive pulmonary disease, congestive heart failure, endocrine system diseases, neurological, psychological diseases, etc.),
* Having a malignant condition,
* Pregnant individuals in the third trimester,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with primary Sjögren's Syndrome according to the American European Consensus Criteria in Hacettepe University, Faculty of Medicine, Rheumatology Department, and volunteers to participate in the study will recruit this study.
  The total number of individuals to be included in the study will be calculated with 80% power and 95% confidence interval with the data obtained after the pilot study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire (BETY-BQ) | baseline
  BETY-BQ consists of the following six subtitles that investigate in detail the biopsychosocial dimensions: pain, functionality and fatigue, mood, sociability, sexuality, and sleep quality. This scale consists of 30 items, scored on a 5-point Likert system. Each question is scored as "No never: 0 Yes rarely: 1 Yes sometimes: 2 Yes often: 3 Yes always: 4" and a total score over 30 items. A higher score indicates a poorer biopsychosocial situation.
Turkish Eating Assessment Tool | baseline
  Turkish Eating Assessment Tool is a survey consisting of 10 questions with a Likert scale between 0 and 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points by finding the sum of the answers given by individuals to each question. A score of 3 or more in the survey is considered abnormal. A score of 16 or above is considered as suspicion of aspiration.
Xerostomia inventory | baseline
  The scale consists of 11 items. Patients will be asked to choose the best response for each item describing their symptoms over the previous two weeks. Responses are scored from 1 to 5 (1: never, 2: rarely, 3: occasionally, 4: fairly often, and 5: very often). The sum of the item scores gives a total score ranging from 11 to 55, and a higher score indicates that the symptoms are more severe.
Multidimensional Fatigue Rating Scale | baseline
  This scale evaluates fatigue with 16 items under 5 subheadings: degree, severity, impact on daily activities, troubles it causes, and fatigue time. The score ranges from 0 (not tired) to 50 (extremely tired).
Hospital Anxiety and Depression Scale (HADS) | baseline
  In this scale consisting of fourteen questions, odd-numbered questions questioning anxiety, and even questions question depression. Options range from 0 to 3, with a higher score indicating a poor emotional state. The cut-off values of the scale were determined as 10 for the anxiety subscale and 7 for the depression subscale.
Test of Mastication and Swallowing Solids | baseline
  In our study, the Test of Masticating and Swallowing Solids (TOMASS) will be used. The test evaluates how many bites the individual takes to eat a biscuit while sitting upright, how many chewing cycles he makes, how many times he swallows it, and how long the total time is from biting to swallowing. Video recording will be taken during the test. The number of bites, number of chewing cycles, number of swallows and total time will be calculated on the video.
Dysphagia limit | baseline
  While evaluating dysphagia, individuals are given 5, 10, 15, 20, 25, 30, 35, 40 and 45 mL volumes of liquid, respectively, with a graduated syringe and are asked to swallow the liquid. The maximum amount of fluid that the thyroid cartilage can swallow during a single movement is determined. The normal dysphagia limit in healthy individuals is more than 20 mL. If a person can swallow 20 mL normally, the dysphagia limit is normal.

SECONDARY OUTCOMES:
Central Sensitization Scale | baseline
  In this scale, which consists of 40 questions and questions the symptoms related to central sensitization, a score above 40 is interpreted as an indicator of central sensitization.
Pain Catastrophizing Scale | baseline
  It is a Likert-type self-assessment scale consisting of 13 items. Each item is scored between 0 and 4 points. The total score ranges from 0 to 52. High scores indicate a high level of catastrophizing. It has 3 subtests: pain magnification (items 6, 7 and 13), rumination (items 8, 9, 10, 11) and helplessness (items 1, 2, 3, 4, 5 and 12).
EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) | baseline
  ESSDAI is a clinical scale that measures disease activity in Sjögren's Syndrome and its items provide objective data consisting of tests applied to patients during routine outpatient clinic check-ups. An ESSDAI score of less than 4 indicates low activity, a score between 5 and 13 indicates moderate activation, and a score of 14 and above indicates high activity.
EULAR Sjögren's Syndrome Patient Reporting Index (ESSPRI) | baseline
  ESSPRI scoring is a symptom severity assessment scale filled out by the patient and used in Sjögren's Syndrome. The patient is asked to express fatigue, pain and dryness complaints with a score between one and ten, and the arithmetic average of the score obtained from these three questions forms the result. An ESSPRI score of less than 5 is considered an acceptable disease state, while a score of 5 or above is considered a sign of high activity.
Primary Sjögren's Syndrome Quality of Life Scale | baseline
  This scale, consisting of twenty-five questions, is divided into two subsections: physical (discomfort and dryness) and psychosocial. Since vaginal dryness, one of the symptoms of SS, was included in the total score, the maximum score was determined as 96 for women and 92 for men. A high score means low health-related quality of life.
Yale Swallow Protocol | baseline
  Protocol has 3 main components: exclusion criteria, short cognitive test and oral mechanism, and drinking 90cc water directly from the glass. Patients who complete step 1 and are not contraindicated for testing proceed to short cognitive testing phase. Patients who pass the short cognitive test and oral mechanism stages can move on to 3th stage, which is drinking 90 cc of water. 90 cc water swallow challenge protocol is a simple assessment that can be used by many qualified healthcare professionals to identify aspiration risk because it is easy to perform, highly reliable, cost-effective, and clinically validated. During test, patient is asked to drink 90 cc of water in consecutive swallows, slowly and continuously but without stopping. Patient is evaluated for signs of i.stopping drinking while drinking, ii.coughing/choking during or immediately after drinking. Patients showing these findings are recorded as 'failing' test.

CONTACTS AND LOCATIONS:
Locations (1):
- Nazli Elif Nacar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No